CLINICAL TRIAL: NCT04855981
Title: Effect of Whole-body Vibration Versus Aerobic Exercise on the Inflammatory Status and Hormonal Parameters in Females With Premenstrual Syndrome
Brief Title: Whole-body Vibration Versus Aerobic Exercise on the Inflammatory Status and Hormonal Parameters Premenstrual Syndrome
Acronym: PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, Principale investigator. al shaymaa shaaban abd el azeim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003183
Record Dates: First submitted 2021-04-07; First posted 2021-04-22 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Premenstrual Syndrome
Keywords: whole body vibration; aerobic exercises; premenstrual syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Exercise; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: whole-body vibration and aerobic exercise
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- whole body vibration (Experimental): the subjects will receive whole-body vibration three times per week for twelve weeks +supplementations
  Interventions: Other: whole body vibration; Other: supplementation
- aerobic exercise (Experimental): the subjects will receive aerobic exercise three times per week for twelve weeks+supplementations
  Interventions: Other: aerobic exercise; Other: supplementation
- supplementations (Active Comparator): the subjects will receive supplementations three times per week for twelve weeks
  Interventions: Other: supplementation

INTERVENTIONS:
Other: whole body vibration — All participants in the WBV group will perform the WBV training on a vibrating device (Confidence Vibration Plate Power Plus, China), which produces a lateral peak-to-peak oscillation. They will stand on the WBV platform with a 150° knee angle during the exposure minute. They started the training with three sets of 1 min separated by a 1-min resting period and vibration amplitude of 1 mm. They will add one set every session until they performed 10 sets of WBV. The frequency started at 20 Hz, which will be increased gradually by 2 Hz every 2 weeks +magnesium (Mg) (250 g) and vitamin B6 supplementation
  Arms: whole body vibration
Other: aerobic exercise — the subjects will receive aerobic exercises+ magnesium (Mg) (250 g) and vitamin B6 supplementation
  Arms: aerobic exercise
Other: supplementation — the subjects will receive magnesium (Mg) (250 g) and vitamin B6 supplementation

SUMMARY:
The purpose of this study is to investigate and compare the effect of whole-body vibration to aerobic exercise on inflammatory status in females with premenstrual syndrome.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) is a complex disorder characterized by moderate to severe symptoms taking place during the luteal phase of the menstrual cycle. It has a negative impact on females' lives, which can affect their relationships, educational efficiency, social activities, and quality of life. Despite previous studies reported that physical exercise improves the symptoms of PMS, the effects of physical exercise on inflammatory status in females with PMS are not clear yet. sixty females allocated to three groups randomly to group (A) that will receive whole-body vibration+supplementation, group (B) that will receive aerobic exercises+supplementation, and group c that will receive supplementation only

ELIGIBILITY:
Inclusion Criteria:

1. Females suffering from PMS (as determined by PMS scale).
2. Their ages will range from 18 to 25 years.
3. Having regular menstrual cycle.

Exclusion Criteria:

1. Smoking.
2. Taking any medications.
3. History of chronic disease.
4. Having any psychiatric or gynecological problems

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
premenstrual symptoms | up to twelve weeks
  The premenstrual syndrome questionnaire also measured the occurrence and severity of two menstrual pain symptoms, including cramp and backache experienced during the first 2 days of the women' last menstrual period. Premenstrual symptoms were scaled as: mild (1); moderate (2); and severe (3). Young women with PMS should experience a premenstrual symptoms score of at least 50% greater than the postmenstrual score

SECONDARY OUTCOMES:
CRP level assessment | up to twelve weeks
  blood sampl a normal reading is less than 10 milligram per liter (mg/L), more than 10 milligram the level of inflammation in body increase.
cortisol level | up to twelve weeks
  When a technician carries out the cortisol level test between 6 a.m. and 8 a.m., the results will typically be within the range of 10-20 micrograms per deciliter (mcg/dL). more than 20 the level of stress increased.
hormonal analysis | up to twelve weeks
  blood sample will be used for assessment the level of progesterone and prolactin. normal level of progesterone less than 0.20 ng/mL and Normal levels of prolactin in females: less than 25 ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Al Shaymaa Shaaban Abd El Azeim, Giza, Egypt